CLINICAL TRIAL: NCT00609245
Title: Effect of Small Changes in Plasma Valproic Acid Concentration on the Photoparoxysmal Response
Brief Title: Effect of Valproic Acid Concentration on Photic Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Bassel Abou-Khalil, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 070849
Record Dates: First submitted 2008-02-01; First posted 2008-02-06 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Photosensitive Epilepsy
Keywords: epilepsy; photosensitive; valproic acid
MeSH Terms: conditions — Epilepsy, Reflex; Epilepsy | interventions — Valproic Acid; Saline Solution; Glucose; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Placebo then Valproic Acid (VPA) (Experimental): all patients will have placebo on day 1 and VPA infusion on day 2
  Interventions: Drug: Valproic Acid; Drug: Placebo

INTERVENTIONS:
Drug: Valproic Acid — The investigators will utilize intravenous sodium valproate at visit 3. Dosage will be individualized to each patient's body weight, age, and hepatic-enzyme-inducing status. Intravenous VPA dose predictions will be based upon population VPA pharmacokinetic parameters (Dutta 2003).
  Other Names: Depacon
Drug: Placebo — Each patient will have a placebo-infusion (with 0.9% NS or D5W) of 12-hour duration at visit 2.
  Other Names: Normal Saline (NS) and 5% Dextrose in water (D5W)

SUMMARY:
We are trying to learn if small changes in the amount of a valproate in the blood (given through an IV) will change the way the brain reacts to flashing lights.

DETAILED DESCRIPTION:
Photosensitive epilepsy is a form of epilepsy that is considered to have a genetic basis in most instances. It is a reflex type of epilepsy. Patients with this condition exhibit epileptic activity patterns (called photoparoxysmal response-PPR) on their EEG during intermittent photic stimulation with certain flash frequencies.

Specific Aims

1. To determine the extent of the pharmacodynamic effect of small changes in total and free VPA concentration via constant infusion of intravenous sodium valproate within the same photosensitive epilepsy patient.
2. To determine the change in total and free VPA concentration required to achieve maximal effect on PPR in patients with photosensitive epilepsy.

Hypothesis

1. Valproic acid (VPA) demonstrates differential pharmacodynamic effect on PPR with small changes in VPA concentration (5-20 mg/L changes in total, or 0.5 to 2 mg/L changes in free VPA) within the same patient. In essence, the VPA concentration-response curve in patients with photosensitive epilepsy is relatively steep.
2. Intravenously-administered VPA will demonstrate a reduction in standard photosensitive range (SPR) or abolition of PPR for at least 80% of patients studied, when the entire range of free VPA concentrations is considered.

Photosensitivity, defined as a PPR on intermittent photic stimulation (IPS), is found in approximately 5% of all epileptic patients. Markedly photosensitive patients are usually sensitive to IPS within clearly defined limits of flash frequency (mostly between 10-30 Hz). This photosensitivity range, the difference between the highest and lowest flash rates that consistently elicit a photoparoxysmal response (PPR), can be used as a quantitative measure of photosensitivity.

Administration of some antiepileptic drugs (AEDS) can diminish or even abolish PPR. With a standard set of tested frequencies, a standard photosensitive range (SPR) can be used to measure drug effect on photosensitivity. Combined with blood level monitoring, the model offers information about actual pharmacodynamic effect as measured with IPS related to the changes in blood levels.

The standardized IPS procedure includes delivery of short (5 second-) trains of flashes. The stimulation starts with the lowest frequencies (which usually do not produce a PPR) only up to the limits of the photosensitivity range (the threshold frequencies for which the patient shows an epileptiform EEG response). After that the stimulation starts again with the highest frequencies (which also do not produce a PPR) down to the frequency that produces a definite PPR.

The photic stimulator will be manually controlled for all stimulations in order to abort the stimulation when a clear PPR is elicited. With all stimulations, there is simultaneous recording of the EEG and direct observation of the patient for clinical changes. With all the safety measures in place, the likelihood of provoking prominent clinical seizures is extremely low.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Aged 15 to 65 years
* Patients with a diagnosis of epilepsy for which they are either taking up two AEDs, not including VPA/divalproex, or no AEDs
* Patients with a reproducible IPS-induced photo-paroxysmal responses of at least 7 SPR-EEG units as measured at two different time points in the day (pm screening Study Visit 1 and am of Visit 2).
* Are in good health (with the exception of epilepsy).
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Patients not exhibiting a photo-paroxysmal-EEG response
* Patients with active psychogenic seizures
* Women who are pregnant or lactating
* Women of reproductive potential who do not agree to use effective birth-control methods during the study and for one week after receiving study drug.
* Patients taking any dosage form of VPA/divalproex within 4 weeks prior to the study
* Patients taking more than two concomitant AEDs
* Patients with any clinically significant laboratory abnormality, which in the opinion of the investigator, will exclude the patient from the study
* Patients who are suffering from active liver disease indicated by abnormal liver function tests greater than three times the upper limit of normal (AST and ALT), patients with porphyria, or patients with a family history of severe hepatic dysfunction
* Patients with a history of alcoholism, drug abuse, or drug addiction (within the past 12 months)
* Patients with a history of sensitivity or allergic reaction to valproate / divalproex
* Patients who have a medical history which would contraindicate sodium valproate (VPA) administration
* Patients who have participated in any other trials involving an investigational product or device within 30 days of screening.
* Patients with clinically significant ECG abnormalities, as judged by the PI, at screening visit
* Patients with such poor intravenous access that the insertion of two intravenous catheters (one for sodium valproate infusion and one, in a contralateral arm vein, for serial blood sampling) for a 12-hour period is not possible.
* Patients who received benzodiazepines within one week of study initiation
* Status epilepticus within one year of screening
* Generalized tonic-clonic seizure within 24 hours of photic stimulation procedure

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bassel Abou-Khalil, MD, Principal Investigator — Vanderbilt University; William Rosenfeld, MD, Principal Investigator — The Comprehensive Epilepsy Care Center for Children & Adults; Dorothee Kasteleijn-Nolst Trenite, MD, PhD, Principal Investigator — The Comprehensive Epilepsy Care Center for Children & Adults
Locations (2):
- United States (2):
  - The Comprehensive Epilepsy Care Center for Children & Adults, Chesterfield, Missouri
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Valproate Infusion: placebo: Each patient will have a placebo-infusion (with 0.9% NS or D5W) of 12-hour duration at visit 2.
  Valproic Acid: The investigators will utilize intravenous sodium valproate at visit 3. Dosage will be individualized to each patient's body weight, age, and hepatic-enzyme-inducing status. Intravenous Na VPA dose predictions will be based upon population VPA pharmacokinetic parameters (Dutta 2003).
Period: Overall Study
Arm/Group | Valproate Infusion
Started | 13
Completed | 12
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Valproate Infusion
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
presence of photoparoxysmal response [Number; unit: participants] | 13

OUTCOME MEASURES:

1. Primary Outcome: Difference in SPR During Placebo and VPA Infusions
Description: standard photosensitive range (SPR) Each participant is exposed to intermittent photic stimulation at 14 predetermined frequencies in order to detect changes in response around typical upper and lower frequency thresholds (e.g., 2 Hz, 5 Hz, 8Hz, 10 Hz, etc.). Each flash frequency that elicits a photosensitive response is considered one "step", and the result is transformed into a metric called the standardized photosensitive range (SPR). The SPR ranges from 0 to 14, where each point represents the number of flash frequencies that elicited a photosensitive response.
Time Frame: At the start of EEG monitoring/drug infusion, and on an hourly basisfor 12 hours
Population: 1 patient did not complete infusion of Valproic Acid due to Adverse Event. This patient was not included in final analysis.
Measure: Mean (Full Range); unit: standard photosensitive range (SPR)
Groups:
- Placebo: Each patient will have a placebo-infusion (with 0.9% NS or D5W) of 12-hour duration.
- Valproic Acid: The investigators will utilize intravenous sodium valproate. Dosage will be individualized to each patient's body weight, age, and hepatic-enzyme-inducing status. Intravenous Na VPA dose predictions will be based upon population VPA pharmacokinetic parameters (Dutta 2003).
Arm/Group | Placebo | Valproic Acid
Number analyzed (Participants) | 12 | 12
standard photosensitive range (SPR) | 15.917 [14.739 to 17.431] | 14.609 [12.903 to 17.124]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.016, ANOVA

ADVERSE EVENTS:
Groups:
- Valproic Acid: Valproic Acid: The investigators will utilize intravenous sodium valproate at visit 3. Dosage will be individualized to each patient's body weight, age, and hepatic-enzyme-inducing status. Intravenous Na VPA dose predictions will be based upon population VPA pharmacokinetic parameters (Dutta 2003).
Arm/Group | Valproic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproic Acid (N=13) | Placebo (N=13)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No